CLINICAL TRIAL: NCT06386068
Title: Interdisciplinary Value-based Cognitive Behavioral Treatment for People with Persistent Whiplash Associated Disorders After Road Traffic Accidents: Protocol for a Multiple Baselines Single-case Experimental Design.
Brief Title: Interdisciplinary Value-based Cognitive Behavioral Treatment for People with Persistent Whiplash Associated Disorders.
Acronym: VALIANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tonny Elmose Andersen, phd., Professor, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2110041
Record Dates: First submitted 2024-01-26; First posted 2024-04-26 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: Whiplash Injuries
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Intervention Model Description: A replicated multiple baselines single-case experimental design with three baseline phases. Baseline randomization into three tiers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baseline phase (Experimental): There are three baseline phases of 1, 2, or 3 weeks to which participants are block-randomized followed by a 10-week intervention phase. Hence, participants are their own case-controls.
  Interventions: Behavioral: Values-based Cognitive Behavioral Therapy (V-CBT)

INTERVENTIONS:
Behavioral: Values-based Cognitive Behavioral Therapy (V-CBT) — The intervention offers a 10-session treatment for chronic Whiplash-Associated Disorder (WAD). The manualized adapted version of value-based cognitive behavioral treatment (V-CBT) is conducted by interdisciplinary teams of psychologists and physiotherapists. The program, based on V-CBT principles, focuses on psychoeducation, fostering self-efficacy, and setting value-based goals in the initial three sessions. The subsequent seven sessions involve physiotherapists trained in V-CBT, addressing psychological, physical, social, and practical barriers hindering engagement in participants' lives. Each session combines psychologically informed themes and supervised exercises, aiming to enhance engagement in values-based activities.

SUMMARY:
The goal of this clinical trial is to address the critical need for effective interventions by developing and testing an interdisciplinary values-based cognitive behavioral therapy (V-CBT) program for individuals with persistent whiplash. The main question it aims to answer are:

* What is the treatment effect of the interdisciplinary values-based cognitive behavioral therapy (V-CBT) program on individuals with persistent whiplash?
* What are the temporal relationships between primary and secondary outcome measures in the context of the V-CBT program?

Participants will undergo a replicated multiple baselines single-case experimental design (SCED). Twelve participants who meet specific eligibility criteria will be block-randomized to a 1, 2, or 3-week baseline phase, serving as their own controls. The intervention involves an interdisciplinary team delivering a manualized adapted V-CBT program over ten sessions, focusing on psychological and physical rehabilitation. Participants will be required to attend these sessions as part of the treatment protocol. Data collection includes daily online self-reports and comprehensive measurements at pre-treatment, post-treatment, and a three-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* have persistent symptoms after a whiplash injury that happened more than 3 months ago
* have pain and disability defined as > 35 % on Neck Disability Index (NDI)
* be 18 years or older
* speak and read Danish

Exclusion Criteria:

* denote headache as the primary problem
* show red flags in the neurological and physiotherapeutic examination such as known or suspected serious spinal pathology, confirmed fracture or dislocation in the neck at the time of injury or signs of nerve root compromise (weakness, reflex changes or sensory loss)
* have had spinal surgery within the past 12 months
* are socially and occupationally unresolved
* have daily significant functional limitations related to other pain conditions
* have severe psychiatric illness
* are pregnant
* are not willing or able to respond to items on a daily basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Value-based living | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on Engaged Living Scale. Scored on a scale from 0 to 10. Higher scores means greater levels of value-based living.
Pain interference | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Three single items focused specifically on general activities, relations with other people, and sleep. Based on Brief Pain Inventory. All three are scored on a scale from 0 to 10. Higher scores means greater levels of pain interference.
Value-based living | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Engaged Living Scale. 16 item scale. Scored on a scale from 1 to 5. Higher total scores indicate greater levels of value-based living.
Pain interference | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Brief Pain Inventory. 7 item scale. Scored on a scale from 0 to 10. Higher total scores indicate greater pain interference.

SECONDARY OUTCOMES:
Pain catastrophizing | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on Daily Pain Catastrophizing Scale). Scored on a scale from 0 to 10. Higher scores means greater levels of pain catastrophizing.
Positive affect | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on previous diary studies. Scored on a scale from 0 to 10. Higher scores means greater levels of positive affect.
Negative affect | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on previous diary studies. Scored on a scale from 0 to 10. Higher scores means greater levels of negative affect.
Stress | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on previous diary studies. Scored on a scale from 0 to 10. Higher scores means greater levels of stress.
Fatigue | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on previous diary studies. Scored on a scale from 0 to 10. Higher scores means greater levels of fatigue.
Pain-related acceptance | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on Chronic Pain Acceptance Questionnaire. Scored on a scale from 0 to 10. Higher scores means greater levels of acceptance.
Pain-related self-efficacy | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on Pain Self-efficacy Questionnaire. Scored on a scale from 0 to 10. Higher scores means greater levels of self-efficacy.
Pain severity | Daily throughout baseline phase (1-3 weeks) and treatment phase (10 weeks).
  Single item measure based on Brief Pain Inventory. Scored on a scale from 0 to 10. Higher scores means greater levels of pain severity.
Neck Disability | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Neck Disability Index. 10 item scale. Scored on a scale from 0 to 5. Higher total scores indicate greater disability.
Depression | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Patient Health Questionnaire (PHQ-9). 9 item scale. Scored on a scale from 0 to 3. Higher total scores indicate greater levels of depression.
Anxiety | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Generalized Anxiety Disorder (GAD-7). 7 items. Scored on a scale from 0 to 3. Higher total scores indicate greater levels of anxiety.
Stress | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Perceived Stress Scale. 10 items. Scored on a 5-point scale. Higher total scores indicate greater levels of stress.
Health-related quality of life | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  EuroQoL-5D-5L. 5 items scored on a 5-point scale and one item scored on a 0 to 100 scale. Higher scores on the first 5 items indicate reduced quality of life and higher scores on the last item indicates greater quality of life.
Pain-related acceptance | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Chronic Pain Acceptance Questionnaire (CPAQ-8). 8 items scored on a scale from 0 to 6. Higher total scores indicate greater levels of acceptance.
Pain-related self-efficacy | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Pain Self-Efficacy Questionnaire. 2 items scored on a scale from 0 to 6. Higher scores indicate greater self-efficacy.
Sleep quality | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Karolinska Sleep Questionnaire. 4 items scores on a scale from 0 to 5. Higher total scores indicates poorer quality of sleep.
Pain severity | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Four 0-10 numeric rating scale (NRS) for worst, mildest, average, and current pain. Scored on a scale from 0 to 10. Higher scores indicate greater levels of pain severity.
Self-perceived improvement | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Global Rating of Change. 1 item scored on a scale from 1 to 15. Higher scores indicate greater level of self-perceived improvement.
Satisfaction with treatment | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Self-developed NRS-item from 0 = not at all satisfied to 10 = completely satisfied.
Pain Disability | Pre-treatment, post-treatment (i.e., within one week from the day of last treatment), 3 months follow-up after treatment completion
  Pain Disability Index. 7 items scored on a scale from 0 to 10. Higher total scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Tonny E Andersen, PhD, Principal Investigator — University of Southern Denmark; Sophie L Ravn, PhD, Study Director — University of Southern Denmark; Anders O Aaby, PhD, Study Director — Specialized Hospital for Polio and Accident Victims
Locations (1):
- Specialized Hospital for Polio and Accident Victims, Rødovre Municipality, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No